CLINICAL TRIAL: NCT05991999
Title: The Effect of Stretching The Pectoralis Major, Sternocleidomastoid, and Iliopsoas Muscles on 800 Meters Swimming Performance in Master Swimmers
Brief Title: The Effect of Stretching of Swimming-related Muscles on 800-meter Swimming Performance in Master Swimmers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYeditepe
Record Dates: First submitted 2023-08-05; First posted 2023-08-15 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Stretch
Keywords: Master swimmer; Swimming; Stretching; 800 meter

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Study Group (Experimental): 800-meter swimming performance tests were administered to all swimmers prior to the measurement. The study group started to do stretch exercises every day for 6 weeks. At the end of six weeks, performance tests and myoton measurements were administered and analyzed for both groups.
  Interventions: Other: Stretching; Other: Training
- The Control Group (Active Comparator): 800-meter swimming performance tests were administered to all swimmers prior to the measurement. The control group just continued their regular training for 6 weeks. At the end of six weeks, performance tests and myoton measurements were administered and analyzed for both groups.
  Interventions: Other: Training

INTERVENTIONS:
Other: Stretching — Master swimmers will be taught iliopsoas, sternocleidomastoid and pectoralis major stretching exercises as stretching exercises. Participants will stretch daily for 3 repetitions, each stretching for 20 seconds.
  Participants will continue their swimming training 2 days a week.
  Arms: The Study Group
Other: Training — Participants continued their swimming training 2 days a week.

SUMMARY:
The study aimed to investigate the effect of stretching the sternocleidomastoid, pectoralis major and iliopsoas muscles on 800 meters freestyle swimming performance in master swimmers.

DETAILED DESCRIPTION:
The benefits of swimming are almost endless. Swimming is important not only as a sport but also for evaluating leisure time, building strength, and recuperating. It even allows some muscles to grow symmetrically and consistently. There is no malfunctioning muscle group in swimming. Even when swimming with minimal effort, one can move with relatively little force and easily. Besides this, it establishes a sense of trust.

Sportive swimming is described as the athlete's ability to complete specific distances in water in the quickest amount of time using freestyle, backstroke, breaststroke, or butterfly strokes. The backstroke technique is performed in supine posture, while the other techniques are swum in facedown, horizontal, and near-horizontal positions. Variable approaches have varied characteristics in terms of body position, leg kick, arm pulling, head position, respiration, and condition.

Biomechanically, our myofascial connections also helps swimmers while they swim. Tightening Superficial Front Line (SFL) causes flexion of the hips and trunk in motion also produces hyperextension at the top of the neck. The large muscles of the pectoralis and latissimus provide the motive force for the large movements of adduction and extension, such as a swimming stroke. Vertical fibers in the fascia on the profound side of the epimysium of the pectoralis major, which does indeed connect from the rectus attachment to the lower part of the fascia colli superficialis (and sternocleidomastoid (SCM)). Lower extremity also coordinates stability while upper part of the body initiates movements between phases İliopsoas starts the hip flexion and is followed up by the rectus femoris initiates knee extension to continue horizontal movement in the water.

Because of the demands of the sport, swimmers have a more rounded forward posture. When the head is forward, the cervical spine is hyperextended, the thoracic spine is in slight flexion, and the lumbar spine is in slight extension, this is known as forward posture. Muscle imbalances in the shoulders are to blame for this forward posture. In the recovery phase of swimming, the scapula must retract and protract along the thoracic wall. The subacromial space reduces with protraction because of the swimmer's adaptation due to sport. Stretching the scapular protractors such as the pectoralis major muscle has been shown to have a considerable impact on the degree of forwarding shoulder posture (FSP) in healthy people. Besides this adaptation also, swimmers with shoulder pain because of more active trigger points can lead to the development of mechanical hypersensitivity compared to ones that do not have any shoulder pain.

As summarized above, swimming athletes generally have a forward posture due to their adaptation to water. In our opinion, this posture may be due to the tension of the anterior group myofascial structures, and releasing the fascia by stretching might affect swimmers' performance. Master swimmers have that adaptation far more compared to young swimmers. Therefore, we can better observe the effects of Sternocleidomastoid, Pectoralis major, and İliopsoas muscle stretching on swimming performance by testing swimmers at distances such as 800 meters.

H0: There is no significant difference between the 800-meter performance measurements of the people in the group that added stretching of specific muscles to their normal training and those in the group that did not add stretching.

H1: There is a significant difference in the 800-meter performance measurements of the group with specific muscle stretching added to their normal training and the people in the group without stretching.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the study voluntarily,
* Participants in ages over 25 years of age,
* Participants must swim at least two days a week.

Exclusion Criteria:

* Presence of chronic disease,
* Participants have undergone surgery in relevant regions in the last 2 years,
* Participants have had injuries in the relevant regions in the last 2 years.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-08-05 (Actual); Primary Completion 2023-10-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
800 Meter Degree test | 6 weeks
  The 800 meter test will be used to evaluate the long-term aerobic metabolic performance of master swimmers.
The MyotonPro - Frequency | 6 weeks
  The tone of muscle is described by frequency of muscle or oscillation frequency (Hz). It evaluates the tone that the muscle is at resting position.
The MyotonPro - Stiffness | 6 weeks
  Stiffness is biomechanical feature of a muscle. It is described by reaction to contraction or forces from outside of tissue that may cause the original form to deteriorate.
The MyotonPro - Decrement | 6 weeks
  The elasticity of a muscle is described by a logarithmic reduction of tissue's normal amplitude. It is more related with the dissipation of mechanical energy that arises between the deformation of the tissue and its recovery. It is a biomechanical feature of tissue that is called as elasticity. When the tissue's decrement is increase, elasticity decreases. There is an opposite proportion among themselves.
The MyotonPro - Relaxation | 6 weeks
  It is the time which is called as Mechanical Stress Relaxation Time (ms) between the deformation of the normal shape of the tissue and its return to its original shape.
The MyotonPro - Creep | 6 weeks
  It is defined as ratio of deterioration and relaxation time of tissue. In case of a continuous stress, tissue regularly stretches over time. This is called as creep.

CONTACTS AND LOCATIONS:
Overall Officials: Şafak Özsönmez, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Ataşehir/İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rittweger J, Kwiet A, Felsenberg D. Physical performance in aging elite athletes--challenging the limits of physiology. J Musculoskelet Neuronal Interact. 2004 Jun;4(2):159-60. No abstract available. PMID 15615117
- [Background] Tanaka H, Seals DR. Endurance exercise performance in Masters athletes: age-associated changes and underlying physiological mechanisms. J Physiol. 2008 Jan 1;586(1):55-63. doi: 10.1113/jphysiol.2007.141879. Epub 2007 Aug 23. PMID 17717011
- [Background] Rubin RT, Rahe RH. Effects of aging in Masters swimmers: 40-year review and suggestions for optimal health benefits. Open Access J Sports Med. 2010 Apr 7;1:39-44. doi: 10.2147/oajsm.s9315. PMID 24198541
- [Background] Batalha NM, Raimundo AM, Tomas-Carus P, Barbosa TM, Silva AJ. Shoulder rotator cuff balance, strength, and endurance in young swimmers during a competitive season. J Strength Cond Res. 2013 Sep;27(9):2562-8. doi: 10.1519/JSC.0b013e31827fd849. PMID 23249824
- [Background] Solem-Bertoft E, Thuomas KA, Westerberg CE. The influence of scapular retraction and protraction on the width of the subacromial space. An MRI study. Clin Orthop Relat Res. 1993 Nov;(296):99-103. PMID 8222458
- [Background] Klingler W, Velders M, Hoppe K, Pedro M, Schleip R. Clinical relevance of fascial tissue and dysfunctions. Curr Pain Headache Rep. 2014;18(8):439. doi: 10.1007/s11916-014-0439-y. PMID 24962403
- [Background] Findley T, Chaudhry H, Stecco A, Roman M. Fascia research--a narrative review. J Bodyw Mov Ther. 2012 Jan;16(1):67-75. doi: 10.1016/j.jbmt.2011.09.004. PMID 22196430
- [Background] Hidalgo-Lozano A, Fernandez-de-las-Penas C, Calderon-Soto C, Domingo-Camara A, Madeleine P, Arroyo-Morales M. Elite swimmers with and without unilateral shoulder pain: mechanical hyperalgesia and active/latent muscle trigger points in neck-shoulder muscles. Scand J Med Sci Sports. 2013 Feb;23(1):66-73. doi: 10.1111/j.1600-0838.2011.01331.x. Epub 2011 May 12. PMID 21564310
- See also: Applications - Myoton. Accessed June 28, 2023 — https://www.myoton.com/applications